CLINICAL TRIAL: NCT02395783
Title: Therapeutic Effects of Maternal Melatonin Administration on Brain Injury and White Matter Disease in Very Preterm Infants
Brief Title: Therapeutic Effects of Maternal Melatonin Administration on Brain Injury and White Matter Disease
Acronym: PREMELIP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P120113
Record Dates: First submitted 2015-03-06; First posted 2015-03-24 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Premature Birth
Keywords: Preterm infants; diagnosis of cerebral white matter injury
MeSH Terms: conditions — Premature Birth | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Melatonin dose1 (Active Comparator): Melatonin 10 µg
  Interventions: Drug: Melatonin 10 µg
- Melatonin dose2 (Active Comparator): Melatonin 20 µg
  Interventions: Drug: Melatonin 20 µg
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin 10 µg — Determine the dose of prenatal administration of melatonin in preterm labor to reduce brain damage in the white matter detected by diffusion tensor imaging (DTI) analysis with spatial statistics (TBSS) to the theoretical term 40 weeks
  Arms: Melatonin dose1
Drug: Melatonin 20 µg — Determine the dose of prenatal administration of melatonin in preterm labor to reduce brain damage in the white matter detected by diffusion tensor imaging (DTI) analysis with spatial statistics (TBSS) to the theoretical term 40 weeks
  Arms: Melatonin dose2
Other: Placebo — Determine the dose of prenatal administration of melatonin in preterm labor to reduce brain damage in the white matter detected by diffusion tensor imaging (DTI) analysis with spatial statistics (TBSS) to the theoretical term 40 weeks
  Arms: Placebo

SUMMARY:
Neurocognitive sequelae observed in preterm represent a major health problem for which there is no preventive treatment approved to date. These effects are the result of a multifactorial brain damage occurring in developing prenatal and perinatal period. Melatonin, the principal hormone secreted by the pineal gland has neuroprotective properties in various experimental animal models of perinatal brain damage level. This hormone readily crosses the placental barrier, its antenatal administration would have a neuroprotective effect in the case of preventive preterm birth before 28 weeks of amenorrhea.

The objective of this study determine the dose of melatonin administered parenterally in prenatal maternal in preterm labor to reduce brain damage in the white matter detected by diffusion tensor imaging (DTI) with statistical spatial analysis (TBSS) to the theoretical term of 40 weeks in children born prematurely.

DETAILED DESCRIPTION:
Neurocognitive sequelae observed in preterm represent a major health problem for which there is no preventive treatment approved to date. These effects are the result of a multifactorial brain damage occurring in developing prenatal and perinatal period. Melatonin, the principal hormone secreted by the pineal gland has neuroprotective properties in various experimental animal models of perinatal brain damage level. This hormone readily crosses the placental barrier, its antenatal administration would have a neuroprotective effect in the case of preventive preterm birth before 28 weeks of gestation.

The objective of this study determine the dose of melatonin administered parenterally in prenatal maternal in preterm labor to reduce brain damage in the white matter detected by diffusion tensor imaging (DTI) with statistical spatial analysis (TBSS) to the theoretical term of 40 weeks in children born prematurely.

Secondary objectives:

* Determine the pharmacokinetics of melatonin administered intravenously in two dosage regimens and after randomization in pregnant women under 28 weeks
* Assess the contribution of antenatal injection of melatonin on the incidence of white matter injury detected by conventional brain MRI
* Assess the contribution of antenatal injection of melatonin on the rate of neurological sequelae at 2 years corrected age, mortality at 28 days of life and at the end of hospitalization.
* Evaluate the adverse effects of melatonin injection

  * Selection criteria (inclusion and non-inclusion)

Inclusion criteria:

* gestational age between 24 weeks + 0 and 27 weeks + 6 days
* Delivery imminent spontaneous defined by cervical dilation greater than or equal to 3 cm and regular contractions, painful (greater than or equal to 2 every 10 minutes) or elective caesarean section.
* maternal age ≥18 years at baseline
* written consent and
* Joining a social security scheme mother and holders of parental authority

Criteria for non-inclusion

Related to the parent criteria:

* Delivery Outborn
* Magnesium Sulphate injection in mother
* Chronic renal and hepatic impairment before pregnancy
* Circumstances of maternal or fetal distress requiring emergency cesarean eclampsia, placental abruption, placenta previa bleeding.

Criteria related to the fetus:

* diagnosis of antenatal malformation Number of subjects required 60 pregnant women between 24 weeks + 0 and 27 weeks + 6 days

  * Search time, duration of participation of each patient Total study duration: 36 months Inclusion period: 12months Duration of participation for a patient 24 months Number of participating centers: 3 Average number of inclusions per month per center: 3
  * Methodology Clinical phase Iib, 3-arms, double-blind randomised controlled trial, multicenter
  * Exams required specifically for research (blood, biopsy ...)
* Treatment: antenatal injection of melatonin ((maximum of 2 doses of 10 mcg or 20 mcg)) against placebo in the delivery room
* Reviews:

  * Determination of plasma melatonin before, after the injection of melatonin (5 minutes, 1 hour, 3 hours, 4 hours after birth) in the mother
  * Determination of plasma melatonin and serotonin in umbilical cord
  * Brain MRI with diffusion tensor sequence (spatial analysis statistiqueTBSS) at 40 weeks • Primary endpoint and secondary endpoints

Primary endpoint:

MRI with diffusion tensor sequence (TBSS analysis).

Standard (s) Secondary Outcome (s):

* Pharmacokinetics of melatonin in the mother
* Determination of plasma melatonin and serotonin in umbilical cord f
* Brain lesions by conventional MRI
* Neurological Evaluation at the age of 2 years by the revised Brunet-test skimped
* Mortality at 28 days of life and at discharge
* Tolerance of melatonin in pregnant women

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 24 weeks + 0 and 27 weeks + 6 days
* Delivery imminent spontaneous defined by cervical dilation greater than or equal to 3 cm and regular contractions, painful (greater than or equal to 2 every 10 minutes) or elective caesarean section.
* maternal age ≥18 years at baseline
* written consent and
* Joining a social security scheme mother and holders of parental authority

Exclusion Criteria:

* Related to the parent criteria:
* Delivery Outborn
* Magnesium Sulphate injection in mother
* Chronic renal and hepatic impairment before pregnancy
* Circumstances of maternal or fetal distress requiring emergency cesarean eclampsia, placental abruption, placenta previa bleeding.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
TBSS analysis | 40 weeks
  The primary endpoint will be the analysis of white matter injury (LSB) at 40 weeks corrected by brain MRI with diffusion tensor sequence (TBSS analysis).

SECONDARY OUTCOMES:
measurement of plasma melatonin levels | before injection of the drug, 5 minutes, 1 hour, 3 hours, 4 hours and 5 hours after injection of the drug
  Pharmacokinetics of melatonin in the mother to determine the dose of Melatonin supplementation in pregnant women (between 24 weeks and 27 weeks + 6days)
Plasma melatonin level | Day 1
  Plasma melatonin level measured in the mother and the newborn at birth (cord blood)
Neurological evaluation (revised Brunet-test) | 2 years
  Neurological evaluation at the age of 2 years by the revised Brunet-test skimped
Mortality | 28 days of life
  Mortality at 28 days of life and at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Biran Valérie, PHD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France